CLINICAL TRIAL: NCT00165087
Title: Treatment of Childhood Acute Lymphoblastic Leukemia
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Terminated by IRB for continuing review
Sponsor: Dana-Farber Cancer Institute (Other)
Collaborators: Boston Children's Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 95-001; NCT00004034 (obsolete NCT alias)
Record Dates: First submitted 2005-09-09; First posted 2005-09-14 (Estimated); Last update posted 2007-12-28 (Estimated); Status verified 2007-12

CONDITIONS: Acute Lymphoblastic Leukemia
Keywords: childhood ALL; standard risk; high risk; infant/high risk
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma | interventions — Asparaginase; Dexrazoxane; Doxorubicin; Radiation

INTERVENTIONS:
Drug: asparaginase (E. Coli)
Drug: asparaginase (Erwina)
Drug: dexrazoxane
Drug: doxorubicin
Procedure: cranial radiation (once daily fractionation)
Procedure: cranial radiation (twice-daily fractionation)
Procedure: Intrathecal chemotherapy without radiation

SUMMARY:
The purpose of this study is to reduce the side-effects and discomfort of anti-leukemia therapy, to attain long-term control of the disease and to hopefully eradicate it.

DETAILED DESCRIPTION:
* Children with acute lymphoblastic leukemia (ALL) are treated somewhat differently depending upon on the relative risk of the leukemia recurring. For this study they are classified into "Standard Risk", "High Risk" and "Infant/High Risk".
* The treatment for patients in the "Standard Risk" and "High Risk" groups consists of three phases of therapy: induction treatment; prevention of brain and spinal cord leukemia (CNS treatment); and intensification/continuation chemotherapy.
* The treatment for patients in the "Infant/High Risk" group consists of four phases of therapy: induction treatment; infant intensification therapy; intensification/continuation chemotherapy; and CNS treatment.
* The induction treatment consists of a combination of chemotherapy drugs whose purpose is to kill all detectable leukemia cells. This process usually requires a least one month and includes six anti-leukemia drugs. These drugs are: vincristine, doxorubicin, methotrexate, cytosine arabinoside, asparaginase and steroids (methylprednisolone or prednisone).
* After the induction phase, "Infant/High Risk" patients will receive a highly intensive month of treatment (infant intensification) . Drugs used during this month include high-dose methotrexate, asparaginase, 6-mercaptopurine and high dose cytosine arabinoside (ARA-C).
* CNS treatment begins during induction therapy but is intensified during the second and third month after diagnosis. Treatment for all patients will include a series of spinal taps with the instillation of anti-leukemia drugs, including cytosine arabinoside and methotrexate and with or without hydrocortisone (depending upon randomization).
* All high risk patients (those in both "High Risk" and "Infant/High Risk") as well as some standard risk patients will receive radiation treatment to the brain. Radiation therapy will either be given in either "conventional" treatments (once daily for 10 days), or "hyperfractionated" treatments (twice daily at half doses for 10 days). Total dose of radiation is 1800 cGy.
* Intensification and continuation therapy, begins 4-5 weeks after diagnosis for "Standard Risk" and "High Risk" groups and 4-5 weeks after infant intensification in "Infant/High Risk" group. This phase of treatment continues until the completion of two years of treatment. Patients in the "Standard Risk" group will receive five anti-leukemia drugs (vincristine, prednisone, methotrexate, asparaginase, and 6-mercaptopurine). Patients in "High Risk" and "Infant/High Risk" will receive six anti-leukemia drugs (vincristine, prednisone, doxorubicin, methotrexate, asparaginase and 6-mercaptopurine).
* All patients will be able to participate in a randomization comparing two types of asparaginase, E.coli and Erwinia. Patients will be randomized to receive either once weekly E.coli or once-weekly Erwinia during the Intensification phase, each given for a total of 20 weeks.
* Patients in the "Standard Risk" group are able to participate in an additional randomization. Standard risk patients will be randomized to receive one of two different regimens designed to prevent central nervous system leukemia, either 1)radiation therapy (given twice daily) with chemotherapy in the spinal fluid every 18 weeks, or 2) intensive chemotherapy in the spinal fluid alone without radiation.
* Patients in the "High Risk" and "Infant/High Risk" groups are able to participate in two randomizations in addition to the asparaginase randomization. The first will be to assess whether the drug dexrazoxane prevents heart damage caused by doxorubicin without affecting risk of relapse. Patients will be randomized to receive either doxorubicin alone or doxorubicin with dexrazoxane during the induction, CNS and intensification phases. The second randomization will compare the relative efficacy and toxicity of different cranial radiation schedules. Patients will be randomized to receive radiation in either once daily or twice daily fractions.
* Blood and bone marrow samples will be collected to learn more about the biology of leukemia. These samples will also be used to test minimal residual disease levels to learn if these levels help predict risk of relapse.
* Quality of life questionnaires will also be performed by the parents of patients, by children over eight, and by the child's clinician.

ELIGIBILITY:
Inclusion Criteria:

* Acute lymphoblastic leukemia, excluding known mature B-cell ALL
* < 18 years of age
* Patients who are leukopheresed or exchanged are eligible for study only after completion of the pheresis or exchange transfusion
* Absence of a t(8,14) (q24; q32), t (8,22), t(2,8)
* Total bilirubin < 1.4mg/dl

Exclusion Criteria:

* Known HIV positive
* Prior steroid therapy within 30 days of diagnosis
* Septic shock
* Ongoing intracranial hemorrhage
* Clinical evidence of CNS or lung leukostasis

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 491
Dates: Start 1996-01; Primary Completion 2006-09 (Actual); Study Completion 2006-09 (Actual)

PRIMARY OUTCOMES:
-To evaluate the efficacy and safety of doxorubicin with or without dexrazoxane
-To determine the efficacy of hyperfractionated radiation plus standard intrathecal chemotherapy compared with intensive intrathecal chemotherapy alone in standard risk patients.
-To compare the relative efficacy and toxicity of E.coli and Erwinia asparaginase
-To compare the relative efficacy and toxicity of cranial radiation delivered in once-daily versus twice-daily fractions in high risk patinets.

SECONDARY OUTCOMES:
-To compare randomized treatment groups using health-related quality of life analyses.

CONTACTS AND LOCATIONS:
Overall Officials: Stephen E. Sallan, MD, Principal Investigator — Dana-Farber Cancer Institute
Locations (10):
- United States (6):
  - Ochsner Clinic, New Orleans, Louisiana
  - Maine Medical Center, Lewiston, Maine
  - Children's Hospital Boston, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - Mt. Sinai Medical Center, New York, New York
  - University of Rochester, Rochester, New York
- Canada (3):
  - McMaster University, Hamilton, Ontario
  - Laval University, Montreal, Quebec
  - Sainte Justine Hosptial, Montreal, Quebec
- San Jorge Children's Hospital, Santurce, Puerto Rico

REFERENCES:
- [Background] Silverman LB, Declerck L, Gelber RD, Dalton VK, Asselin BL, Barr RD, Clavell LA, Hurwitz CA, Moghrabi A, Samson Y, Schorin MA, Lipton JM, Cohen HJ, Sallan SE. Results of Dana-Farber Cancer Institute Consortium protocols for children with newly diagnosed acute lymphoblastic leukemia (1981-1995). Leukemia. 2000 Dec;14(12):2247-56. doi: 10.1038/sj.leu.2401980. PMID 11187916
- [Background] Silverman LB, Gelber RD, Dalton VK, Asselin BL, Barr RD, Clavell LA, Hurwitz CA, Moghrabi A, Samson Y, Schorin MA, Arkin S, Declerck L, Cohen HJ, Sallan SE. Improved outcome for children with acute lymphoblastic leukemia: results of Dana-Farber Consortium Protocol 91-01. Blood. 2001 Mar 1;97(5):1211-8. doi: 10.1182/blood.v97.5.1211. PMID 11222362
- [Background] Goldberg JM, Silverman LB, Levy DE, Dalton VK, Gelber RD, Lehmann L, Cohen HJ, Sallan SE, Asselin BL. Childhood T-cell acute lymphoblastic leukemia: the Dana-Farber Cancer Institute acute lymphoblastic leukemia consortium experience. J Clin Oncol. 2003 Oct 1;21(19):3616-22. doi: 10.1200/JCO.2003.10.116. PMID 14512392
- [Result] Lipshultz SE, Rifai N, Dalton VM, Levy DE, Silverman LB, Lipsitz SR, Colan SD, Asselin BL, Barr RD, Clavell LA, Hurwitz CA, Moghrabi A, Samson Y, Schorin MA, Gelber RD, Sallan SE. The effect of dexrazoxane on myocardial injury in doxorubicin-treated children with acute lymphoblastic leukemia. N Engl J Med. 2004 Jul 8;351(2):145-53. doi: 10.1056/NEJMoa035153. PMID 15247354
- [Result] Waber DP, Silverman LB, Catania L, Mautz W, Rue M, Gelber RD, Levy DE, Goldwasser MA, Adams H, Dufresne A, Metzger V, Romero I, Tarbell NJ, Dalton VK, Sallan SE. Outcomes of a randomized trial of hyperfractionated cranial radiation therapy for treatment of high-risk acute lymphoblastic leukemia: therapeutic efficacy and neurotoxicity. J Clin Oncol. 2004 Jul 1;22(13):2701-7. doi: 10.1200/JCO.2004.10.173. PMID 15226337
- [Derived] Burns MA, Place AE, Stevenson KE, Gutierrez A, Forrest S, Pikman Y, Vrooman LM, Harris MH, Hunt SK, O'Brien JE, Asselin BL, Athale UH, Clavell LA, Cole PD, Gennarini LM, Kahn JM, Kelly KM, Laverdiere C, Leclerc JM, Michon B, Schorin MA, Sulis ML, Welch JJG, Neuberg DS, Sallan SE, Silverman LB. Identification of prognostic factors in childhood T-cell acute lymphoblastic leukemia: Results from DFCI ALL Consortium Protocols 05-001 and 11-001. Pediatr Blood Cancer. 2021 Jan;68(1):e28719. doi: 10.1002/pbc.28719. Epub 2020 Oct 7. PMID 33026184
- [Derived] Lipshultz SE, Scully RE, Lipsitz SR, Sallan SE, Silverman LB, Miller TL, Barry EV, Asselin BL, Athale U, Clavell LA, Larsen E, Moghrabi A, Samson Y, Michon B, Schorin MA, Cohen HJ, Neuberg DS, Orav EJ, Colan SD. Assessment of dexrazoxane as a cardioprotectant in doxorubicin-treated children with high-risk acute lymphoblastic leukaemia: long-term follow-up of a prospective, randomised, multicentre trial. Lancet Oncol. 2010 Oct;11(10):950-61. doi: 10.1016/S1470-2045(10)70204-7. Epub 2010 Sep 16. PMID 20850381